CLINICAL TRIAL: NCT02045576
Title: Positional Therapy With the Sleep Position Trainer Versus Oral Appliance Therapy in Patients With Position Dependent Obstructive Sleep Apnea; A Randomised Controlled Trial
Brief Title: RCT: Oral Appliance Therapy and Sleep Position Trainer in Patients With Position Dependant Obstructive Sleep Apnea
Acronym: POSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: St. Lucas Andreas Ziekenhuis Hospital (Other)
Responsible Party: Principal Investigator, M.H.T. de Ruiter, Resident/PhD student, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POSA
Record Dates: First submitted 2013-11-26; First posted 2014-01-27 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Obstructive Sleep Apnea; Sleep Position Trainer; Oral Appliance Therapy
Keywords: Obstructive Sleep Apnea; sleep position trainer; oral appliance therapy; mandibular advancement device or splint
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleep position trainer (Experimental): Nightbalance
  Interventions: Device: sleep position trainer
- Oral Appliance Therapy (Active Comparator): Somnodent
  Interventions: Device: Oral Appliance Therapy

INTERVENTIONS:
Device: sleep position trainer
  Other Names: Nightbalance
  Arms: Sleep position trainer
Device: Oral Appliance Therapy
  Other Names: Somnodent
  Arms: Oral Appliance Therapy

SUMMARY:
SUMMARY Rationale: Fifty-six percent of patients with Obstructive Sleep Apnea (OSA) are position dependent, defined as having an AHI, which is at least twice as high in supine sleeping position compared to the AHI during sleep in other positions. Standard therapy for patients having mild or moderate POSA is treatment with an Oral Appliance Trainer (OAT). Recently a new device Sleep Position Trainer (SPT) is been introduced especially for patients with POSA.

Objective: To compare the effect of positional therapy with the SPT versus OAT on polysomnographic (PSG) parameters, to evaluate the compliance and measuring the possible learning effect that might occur with POSA patients using the SPT for positional therapy over a long term.

Study design: Randomised controlled trial Study population: The participants of the research will be recruited from the departments of Otolaryngology and Clinical Neurophysiology, Saint Lucas Andreas Hospital, Amsterdam, the Netherlands.

Participants will be males or females older than 18 years with diagnosis of positional OSA.

Intervention: The SPT is a sensor positioned in an elastic band attached around the body. The SPT measures the body position and vibrates when the patient lies in supine position. Oral appliance therapy (OAT) is an intra-oral prosthesis, which holds the mandible in a protrusive position. Because of this position more pharyngeal space will be available and the AHI will decrease. After randomisation the first group (n=45) will sleep for a period of 90 +/- 2 days with the SPT every night. The second group (n=45) will also sleep for a period of 90 +/- 2 days only with OAT. After this period the PSG is repeated. Long- term outcome in AHI is measured by repeating the PSG after 1 year. Main study parameters/ endpoints: Primary endpoints; reduction of PSG parameters, in particular AHI, AI, HI, DI, reduction of % of sleeping supine sleep position, without disturbance of the sleep quality.

Secondary endpoints: Outcome of Quality of Life questionnaires; EQ-5D, ESS, FOSQ and MFIQ.

Compliance and learning effect will also be evaluated for the time period of 3 and 12 months. Finally cardiovascular parameters like blood pressure, pulse rate and BMI/neck circumference will be assessed.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risks for patients participating in this study are negligible. Inconveniences of the SPT can be discomfort caused by irritation of the band, difficulties with an increased sleeping period on the side or difficulties sleeping with the SPT. This can be compensated by the expected improvement of sleep quality caused by the therapy. Possible side effects of OAT may be discomfort in the jaw, sensitivity of the teeth and a dry mouth. Withdrawing from this therapy means immediate relief of inconveniences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older.
* Ability to speak, read and write Dutch.
* Ability to follow up.
* Ability to use a computer with internet connection and windows-software for uploading data and online questionnaires.
* Diagnosis with symptomatic mild or moderate OSA (5 < AHI < 30).
* Diagnosis of 10 to 90% supine position during the night.
* AHI supine is >2 times as high as AHI non-supine.
* Expected to maintain current lifestyle (sports, medicine, diet etc.).

Exclusion Criteria:

* Many dental problems; insufficient teeth for wearing OAT.
* Medication used/ related to sleeping disorders.
* Central Sleep Apnoea Syndrome.
* Night or shifting work.
* Severe chronic heart failure.
* Medical history of known causes of tiredness by day or severe sleep disruption (insomnia, PLMS, Narcolepsy).
* Seizure disorder.
* Known medical history of mental retardation, memory disorders or psychiatric disorders.
* Patients with old type of pacemakers (It is possible that old types of peacemakers are not compatible with the electromagnetic radiation of the electronics of the SPT).
* Shoulder, neck and back complaints.
* Reversible morphological upper airway abnormalities (e.g. enlarged tonsils).
* Inability to provide informed consent.
* Simultaneous use of other treatment modalities to treat OSA.
* Previous treatment for OSA with OAT or SPT
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Efficacy in reducing the mean AHI | 12 months
  Apnoea Hypopnoea Index (AHI)

SECONDARY OUTCOMES:
effectiveness in quality of life | 3, 6, 9 and 12 months
  Outcomes in QoL- questionnaires:
  EQ-5D, Epworth Sleeping Scale (ESS), Functional Outcome Sleep Questionnaire (FOSQ), Mandibular Function Impairment Questionnaire (MFIQ).
Compliance | 3, 6, 9, 12 months
  Actual wearing time in minutes per night
Cardiovascular parameters | 3, 6, 9, 12 months
  Blood pressure
Cardiovascular parameters | 3, 6, 9 and 12 months
  Pulse

OTHER OUTCOMES:
Body Mass Index | Baseline, 3, 6, 9, 12 months
Neck circumference | Baseline, 3, 6, 9, 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - St Lucas Andreas Hospital, Amsterdam

REFERENCES:
- [Derived] de Ruiter MHT, Benoist LBL, de Vries N, de Lange J. Durability of treatment effects of the Sleep Position Trainer versus oral appliance therapy in positional OSA: 12-month follow-up of a randomized controlled trial. Sleep Breath. 2018 May;22(2):441-450. doi: 10.1007/s11325-017-1568-4. Epub 2017 Sep 15. PMID 28913630
- [Derived] Benoist L, de Ruiter M, de Lange J, de Vries N. A randomized, controlled trial of positional therapy versus oral appliance therapy for position-dependent sleep apnea. Sleep Med. 2017 Jun;34:109-117. doi: 10.1016/j.sleep.2017.01.024. Epub 2017 Mar 27. PMID 28522078